CLINICAL TRIAL: NCT05122559
Title: Randomized Controlled Trial of N-acetyl Cysteine as a Neuroprotective Agent in Progressive Multiple Sclerosis
Brief Title: Neuroprotection With N-acetyl Cysteine for Patients With Progressive Multiple Sclerosis
Acronym: NACPMS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emmanuelle Waubant, MD PhD (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Emmanuelle Waubant, MD PhD, Professor, Neurology UCSF Weill Institute for Neurosciences, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P0549747
Record Dates: First submitted 2021-11-08; First posted 2021-11-16 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Primary Progressive; Multiple Sclerosis, Secondary Progressive
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetyl cysteine (Active Comparator): N-acetyl cysteine (NAC) 1200mg t.i.d.
  Interventions: Drug: N-acetyl cysteine
- Placebo (Placebo Comparator): Placebo 1200mg t.i.d.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetyl cysteine — N-acetyl cysteine (NAC) is a Glutathione (GSH) precursor with antioxidant properties which make it relevant for neuroprotection.
  Other Names: NAC
  Arms: N-acetyl cysteine
Drug: Placebo — Lactose Monohydrate, USP (100%), magnesium stearate, silicon dioxide NF
  Arms: Placebo

SUMMARY:
This study evaluates the effectiveness of N-acetyl cysteine (NAC) in the treatment of progressive multiple sclerosis. Half of the patients will receive NAC, while the other half will receive a placebo.

ELIGIBILITY:
Inclusion Criteria:

* - 40-70 (inclusive) years in age,
* meet 2017 McDonald criteria (Thompson 2018),
* patients with primary or secondary progressive MS (Thompson 2018),
* at least 2 years since progressive symptom onset,
* evidence of clinical changes over the previous 2 years unrelated to relapses: increased EDSS or 20% slowing on 25-foot walk, change of ambulatory support, cognitive change documented on cognitive testing. Progression defined by patients in terms of ambulation perimeter or type of support to ambulate are acceptable if aforementioned physician-based measure changes are not available.
* EDSS score 3.0 to 7.0 (inclusive),
* can be on a stable disease-modifying treatment initiated > 3 months prior to screening,
* can be on stable doses of dalfampridine initiated at least one month before screening.

Exclusion Criteria:

* - MS relapses in the previous 6 months
* oral glucocorticosteroid treatment within the prior 3 months
* patient with issues undergoing MRI scans
* pregnancy or breastfeeding
* women of child-bearing potential not able to utilize an effective form of contraception for the duration of the study
* history of bleeding disorders
* active gastrointestinal ulcers
* abnormal liver function testing (aminotransferase (AST) or alanine aminotransferase (ALT) >2 times upper limit of normal)
* current treatment for active malignancy or metastatic malignancy treated in the past year
* alcohol or substance use disorder
* allergy to NAC
* planned surgery or move within 15 months
* use of medications/supplements with antioxidant properties (including over-the-counter NAC)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 15 months
  Number of adverse events recorded by system, severity, and by relationship to treatment arm.
Effect of NAC on on progression of brain, thalamic and cervical cord atrophy | 15 months
  The primary endpoint is brain, thalamic and cord atrophy measured by brain and cervical spine MRI at month 3 and month 15.

SECONDARY OUTCOMES:
Clinical effects of NAC | 15 months
  Clinical effects in MS as measured by the 9-HPT, 25-foot walk, symbol digit modalities test (SDMT).

OTHER OUTCOMES:
Effect of NAC on progression of MS | 15 months
  Monitoring progression using imaging metrics and changes captured by a wearable multi-sensor device.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schoeps VA, Graves JS, Stern WA, Zhang L, Nourbakhsh B, Mowry EM, Henry RG, Waubant E. N-Acetyl Cysteine as a Neuroprotective Agent in Progressive Multiple Sclerosis (NACPMS) trial: Study protocol for a randomized, double-blind, placebo-controlled add-on phase 2 trial. Contemp Clin Trials. 2022 Nov;122:106941. doi: 10.1016/j.cct.2022.106941. Epub 2022 Sep 28. PMID 36182028